CLINICAL TRIAL: NCT02249559
Title: Pilot Study Evaluating Safety of Unilateral Gamma Knife Subthalamotomy for Parkinson's Disease
Acronym: GKSTN
Status: Terminated | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 14-00902
Record Dates: First submitted 2014-09-12; First posted 2014-09-25 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Parkinsons Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- GK subthalamotomy: Evaluate the safety and efficacy of unilateral GK subthalamotomy for PD in patients deemed poor candidates for DBS.

SUMMARY:
This is a pilot study to evaluate the safety and efficacy of unilateral gamma knife subthalamotomy for Parkinson's disease in patients deemed poor candidates for deep brain stimulation.

DETAILED DESCRIPTION:
The goal of the study is to enroll 20 subjects who could benefit from unilateral subthalamotomy due to the presence of unilateral rigidity, tremor, bradykinesia and/or dyskinesias (as opposed to axial symptoms such as walking) but who are suboptimal candidates for deep brain stimulation (DBS) because of advanced age (>74), medical comorbidities precluding surgery, or patient aversion to DBS, and who show more than 30% improvement in Unified Parkinson's Disease Rating Scale (UPDRS) score in the ON versus OFF medication state.

Secondary objectives will focus on the efficacy of Gamma Knife (GK) subthalamotomy for Parkinson's disease (PD), as determined by changes in the patient's clinical status and any improvement following the treatment. A full neurologic exam as well as a screen for depression will be administered at every postoperative visit. The patient's neurologic function will be assessed with a full neurological examination and objectively quantified using the UPDRS focusing on the contralateral side, as well as overall UPDRS.

The clinician will complete a Clinical Global Impression (CGI) and Mini-Mental State Examination (MMSE) at each visit to record overall impression of the patient's disease progression and severity, and to evaluate cognitive function. Pre- and post-treatment assessment of the Levodopa Equivalent Daily Dose (LEDD) (quantification of medication regimen in levodopa equivalents) will be obtained and recorded to evaluated the efficacy of gamma knife subthalamotomy (GKS) as a treatment for Parkinson's disease (PD). A Parkinson's Disease Questionnaire-39 (PDQ-39) to determine the patient's independence and quality of life will be filled out at each visit. Finally, the patient will complete a Beck Depression Inventory at each clinic visit to monitor for development or progression of depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Otherwise appropriate DBS candidates but deemed suboptimal for DBS on account of one or more of the following:

   * advanced age greater than 74 years of age
   * medical comorbidities

     * need for continual anticoagulation
     * poor candidates for general anesthesia based on cardiac, hepatic ,renal or pulmonary status
     * high infection risk if internal DBS device hardware is placed (ie. Poor diabetes mellitus control)
   * patient aversion to DBS
2. Patients with asymmetric disease symptoms including:

   * rigidity
   * tremor
   * bradykinesia
   * dyskinesia
3. More than 30% improvement in UPDRS score in ON versus OFF medication state, except:

   * in the presence of disabling contralateral dyskinesias/dystonia limiting dose tolerance
   * tremors that are medically refractory
4. Patients who are on a stable medication regimen and demonstrating stable disease symptoms (absence of significant improvement or deterioration) for at least 3 months at the time of GKS, as determined by review of medical record
5. MMSE score greater than or equal to 26

Exclusion Criteria:

* Patients with prominent axial symptoms including postural instability and gait disturbances, defined as a score of 3 or greater on Questions 28, 29 & 30 on the UPDRS
* Patients whose symptoms do not improve by more than 30% in UPDRS score with medication, unless patient experiences dose-limiting side effects
* The presence of dementia or inability to provide informed consent for participation in the study, as determined by a mini-mental status examination score below 25
* Patients who have had prior brain radiation
* Patients with improvement and satisfactory symptom management will not be offered this procedure. We will only include patients without satisfactory symptom management.

Min Age: 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Safety of performing GK lesions in the Subthalamic Nucleus (STN) for PD patients | 12 months
  * Safety of GK subthalamotomy in the management of PD as measured by stable findings on neurologic exam at each clinic visit (hemiballismus, dyskinesias, sensory changes) and the absence of Serious Adverse Events (SAE) attributable to treatment.
  * Because this study does not have a control group, we will compare the non-inferiority of GK subthalamotomy to published outcomes in PD patients undergoing other forms of management.

SECONDARY OUTCOMES:
Efficacy of GK subthalamotomy for PD | 12 months
  To be determined by changes in the patient's clinical status and any improvement following the treatment.
  * Neurologic function as determined by UPDRS, MMSE, neurologic exam results, CGI assessment and LEDD score.
  * Quality of life, as determined by PDQ-39 score and Beck's Depression Inventory (BDI) score.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Kondziolka, MD, Principal Investigator — NYU MEDICAL CENTER
Locations (1):
- NYU Medical Center, New York, New York, United States